CLINICAL TRIAL: NCT02645890
Title: A Randomized, Open-label, Oral Single Dosing, Two-way Crossover Clinical Trial to Evaluate the Safety and Pharmacokinetic Profiles of CKD-397 in Healthy Male Subjects
Brief Title: Study to Compare the Safety and Pharmacokinetics of CKD-397
Acronym: CKD-397
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 150BPH15022
Record Dates: First submitted 2015-12-21; First posted 2016-01-05 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia; Healthy Male Volunteer; Tamsulosin; Tadalafil
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CKD-397 (Active Comparator): Tadalafil/ Tamsulosin Fixed dose combination
  Interventions: Drug: CKD-397
- TD+TM (Experimental): Tadalafil/ Tamsulosin Coadministration
  Interventions: Drug: TD+TM

INTERVENTIONS:
Drug: CKD-397 — Arm A:Tamsulosin/ Tadalafil Fixed dose combination
  Other Names: Arm A
  Arms: CKD-397
Drug: TD+TM — Arm B: Tamsulosin/ Tadalafil Coadministration
  Other Names: Arm B
  Arms: TD+TM

SUMMARY:
The purpose of this study is to compare the safety and pharmacokinetics profiles of CKD-397 in healthy male volunteers.

DETAILED DESCRIPTION:
A randomized, open-label, oral single dosing, two-way crossover clinical trial to evaluate the safety and pharmacokinetic profiles of CKD-397 in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

1. More than 19 years in Healthy male volunteer
2. Body weight ≥ 55kg and in the range of calculated BMI 17.5 to 30.5kg/m2
3. Subject who signed on an informed consent form willingly

Exclusion Criteria:

1. Clinically significant disease with hematological, nephrological, respiratory, gastrointestinal, urogenital, cardiovascular, psychiatric, neurologic system and allergic disease (except for non-symptom seasonal allergy)
2. Gastrointestinal disease(esophageal achalasia, esophagus stenosis, crohn's disease) or gastrointestinal surgery(except for appendectomy or herniotomy)
3. Aspartate aminotransferase, Alanine aminotransferase > 2 X upper limit of normal range or eGFR which is calculated by MDRD(Modification of diet in renal disease) < 60mL/min/1.73m2
4. Continuously taking excessive alcohol(>210g/week) within 6 months before screening
5. Have received any other investigational drug within 3 months prior to the first dosing
6. Sitting systolic blood pressure ≤ 100mmHg or ≥ 150mmHg, sitting diastolic blood pressure ≤ 60mmHg or ≥ 100mmHg
7. Subject with orthostatic hypotension
8. The history of drug abuse or drug abuse showed a positive for urine drug test
9. Subject who takes inducers or inhibitors of drug metabolizing enzyme within 30 days
10. Cigarette ≥ 20 cigarettes a day for recent 3 months and Subject who cannot stop smoking during clinical trial participation
11. Subject who takes ethical drug or herbal medicine within 2 weeks or over-the-counter drug or vitamins within 1 week
12. Whole blood donation within 2 months or component blood donation within 1 month or blood transfusion within 1 month prior to the first dosing
13. Subject who can increase risk due to clinical test and administration of drugs or has severe grade / chronic medical, mental condition or abnormal laboratory result that may interfere with the analysis of test results.
14. Subject with taking any forms of organic nitrate periodically and/or intermittently.
15. Subject with known hereditary degenerative retinal disease including retinitis pigmentosa.
16. Subject with serious history of hypersensitivity to investigational product (including Tadalafil and Tamsulosin) and other medicine (aspirin, antibiotics and so on)
17. Subject who lost sight of one eye by non-arteritic anterior ischemic optic neuropathy (NAION, non-arteritic anterior ischemic optic neuropathy).
18. Subject with genetic problems such as galactose intolerance, fructose intolerance, lapp lactase deficiency, glucose-galactose malabsorption or sucrase-isomaltase insufficiency
19. Subject who planned pregnancy during clinical trial and doesn't use trustworthy contraception
20. Subjects who is not able to comply with guidelines described in the protocol.
21. An impossible one who participants in clinical trials by investigator's decision including laboratory test result or another reason

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
AUC0-t of Tadalafil/ Tamsulosin | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours

SECONDARY OUTCOMES:
Cmax of Tadalafil/ Tamsulosin | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
AUCinf of Tadalafil/ Tamsulosin | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
Tmax of Tadalafil/ Tamsulosin | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
t1/2 of Tadalafil/ Tamsulosin | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
CL/F of Tadalafil/ Tamsulosin | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
Vd/F of Tadalafil/ Tamsulosin | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Min Kyu Park, MD, PhD, Principal Investigator — 9F, DongA University Hospital Department of clinical pharmacology, #26, Daechingongwon-ro, seo-gu, busan, 49201, KOREA
Locations (1):
- Dong A University Hospital, Seo-gu, Busan, South Korea